CLINICAL TRIAL: NCT04524715
Title: Low-Level Laser Therapy Treatment of Lung Inflammation in COVID-19 Patients
Brief Title: LLLT Treatment of Lung Inflammation in COVID-19
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Based upon feedback from IRB.
Sponsor: Ward Photonics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CP19-02
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Blinded before and after comparison of COVID-19 patients treated with a red-light LLLT therapy in addition to standard treatment measures compared to a control group receiving only standard treatment measures.
Who Masked: Participant
Masking Description: All participants undergo LLLT treatment; however, the active group receives LED light in the red and IR range while the placebo group is told they are receiving IR light not visible to naked eye. All participants continue receiving standard treatments for COVID19 symptoms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Treatment Group (Experimental): LLLT Treatment using an UltraSlim red/IR LED device along with all standard treatment measures for COVID19.
  Interventions: Device: Non-invasive red LLLT treatment to chest of patient.
- Control Group (Sham Comparator): Treatment using a Sham comparator along with all standard treatment measures for COVID19.
  Interventions: Device: Sham Device Treatment

INTERVENTIONS:
Device: Non-invasive red LLLT treatment to chest of patient. — Expose patient to LLLT light while lying on their back, elevated at an angle of approximately 45 degrees from horizontal. Position light over the patient's chest at a 33-degree bias to their right and left sides for 20 minutes each side respectively.
  Arms: Active Treatment Group
Device: Sham Device Treatment — Expose patient to sham device while lying on their back, elevated at an angle of approximately 45 degrees from horizontal. Position light over the patient's chest at a 33-degree bias to their right and left sides for 20 minutes each side respectively.
  Arms: Control Group

SUMMARY:
To determine if a reduction of pneumonic inflammation occurs after treatment with Low-Level Laser Therapy (LLLT) applying red-light technology in the respiratory system of COVID-19 patients suffering from acute viral pneumonia.

DETAILED DESCRIPTION:
This clinical trial is a blinded before and after comparison of the effect on patients treated with a red-light LLLT therapy for acute lung inflammation as a result of COVID-19 infection. Patients are enrolled to undergo LLLT therapy in addition to all standard ongoing therapies for COVID-19.

Outcomes for patients receiving LLLT in addition to their standard care (the treatment group) are compared to the group receiving only standard therapy for COVID-19 (control group). Effects of LLLT treatment are measured immediately following treatment, and outcome measurements are compared to the pre-treatment baseline.

ELIGIBILITY:
Inclusion Criteria:

* Participant is diagnosed with COVID-19.
* Study participant is 18 years of age or older.
* Patient exhibiting moderate-to-acute respiratory distress.

Exclusion Criteria:

* Photosensitive condition or medication.
* Active chemotherapy treatment or other cancer treatment.
* Autoimmune Disorder.
* Pregnant, possibly pregnant or planning pregnancy prior to the end of study participation.
* Developmental disability or cognitive impairment that, in the opinion of the investigator, would preclude adequate comprehension of the informed consent form and/or ability to record the necessary study measurements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-31 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Inflammation of the lungs - O2 | 10 days
  Change in inflammation of the lungs as measured by O2 saturation levels
Inflammation of the lungs - CRP | 10 days
  Change in inflammation of the lungs as measured by C-Reactive Protein (CRP) Test
Inflammation of the lungs - IL6 | 10 days
  Change in inflammation of the lungs as measured by IL-6 Levels

CONTACTS AND LOCATIONS:
Overall Officials: Rober H Burke, MD, Principal Investigator — Michigan Center for Cosmetic Surgery
Locations (1):
- Wellness Junction, Millsboro, Delaware, United States

IPD SHARING:
Plan to Share IPD: No
This investigational study is exploratory in nature. The primary endpoint is most descriptive in statistical terms of whether the active patient group had significantly better outcomes than the control group. Individual patient data may be explored at a later date to determine related factors such as patient demographics, comorbidities, or other evidence of compounding variables.

REFERENCES:
- [Background] Hamblin MR. Mechanisms and applications of the anti-inflammatory effects of photobiomodulation. AIMS Biophys. 2017;4(3):337-361. doi: 10.3934/biophy.2017.3.337. Epub 2017 May 19. PMID 28748217
- [Background] Rigonato-Oliveira NC, de Brito AA, Vitoretti LB, de Cunha Moraes G, Goncalves T, Herculano KZ, Alves CE, Lino-Dos-Santos-Franco A, Aimbire F, Vieira RP, Ligeiro de Oliveira AP. Effect of Low-Level Laser Therapy (LLLT) in Pulmonary Inflammation in Asthma Induced by House Dust Mite (HDM): Dosimetry Study. Int J Inflam. 2019 Mar 21;2019:3945496. doi: 10.1155/2019/3945496. eCollection 2019. PMID 31015955
- [Background] Gattinoni L, Chiumello D, Caironi P, Busana M, Romitti F, Brazzi L, Camporota L. COVID-19 pneumonia: different respiratory treatments for different phenotypes? Intensive Care Med. 2020 Jun;46(6):1099-1102. doi: 10.1007/s00134-020-06033-2. Epub 2020 Apr 14. No abstract available. PMID 32291463
- [Background] de Lima FM, Villaverde AB, Albertini R, Correa JC, Carvalho RL, Munin E, Araujo T, Silva JA, Aimbire F. Dual Effect of low-level laser therapy (LLLT) on the acute lung inflammation induced by intestinal ischemia and reperfusion: Action on anti- and pro-inflammatory cytokines. Lasers Surg Med. 2011 Jul;43(5):410-20. doi: 10.1002/lsm.21053. PMID 21674546
- [Background] Chen S, Li Y, Zheng Z, Luo Q, Chen R. The analysis of components that lead to increased work of breathing in chronic obstructive pulmonary disease patients. J Thorac Dis. 2016 Aug;8(8):2212-8. doi: 10.21037/jtd.2016.08.01. PMID 27621878
- [Background] Miranda da Silva C, Peres Leal M, Brochetti RA, Braga T, Vitoretti LB, Saraiva Camara NO, Damazo AS, Ligeiro-de-Oliveira AP, Chavantes MC, Lino-Dos-Santos-Franco A. Low Level Laser Therapy Reduces the Development of Lung Inflammation Induced by Formaldehyde Exposure. PLoS One. 2015 Nov 16;10(11):e0142816. doi: 10.1371/journal.pone.0142816. eCollection 2015. PMID 26569396
- [Background] da Cunha Moraes G, Vitoretti LB, de Brito AA, Alves CE, de Oliveira NCR, Dos Santos Dias A, Matos YST, Oliveira-Junior MC, Oliveira LVF, da Palma RK, Candeo LC, Lino-Dos-Santos-Franco A, Horliana ACRT, Gimenes Junior JA, Aimbire F, Vieira RP, Ligeiro-de-Oliveira AP. Low-Level Laser Therapy Reduces Lung Inflammation in an Experimental Model of Chronic Obstructive Pulmonary Disease Involving P2X7 Receptor. Oxid Med Cell Longev. 2018 Mar 4;2018:6798238. doi: 10.1155/2018/6798238. eCollection 2018. PMID 29686745
- [Background] Oliveira MC Jr, Greiffo FR, Rigonato-Oliveira NC, Custodio RW, Silva VR, Damaceno-Rodrigues NR, Almeida FM, Albertini R, Lopes-Martins RA, de Oliveira LV, de Carvalho Pde T, Ligeiro de Oliveira AP, Leal EC Jr, Vieira RP. Low level laser therapy reduces acute lung inflammation in a model of pulmonary and extrapulmonary LPS-induced ARDS. J Photochem Photobiol B. 2014 May 5;134:57-63. doi: 10.1016/j.jphotobiol.2014.03.021. Epub 2014 Apr 4. PMID 24792475